CLINICAL TRIAL: NCT02831166
Title: A Randomized Comparison Between Transfemoral Approach With Vascular Closure Device Versus Transradial Approach in Primary Percutaneous Coronary Intervention
Brief Title: Vascular Closure Device Versus Transradial Approach in Primary Percutaneous Coronary Intervention
Acronym: ARISE-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Irmandade Santa Casa Misericórdia Marília (Other)
Responsible Party: Principal Investigator, Pedro Beraldo de Andrade, MD, phD, Irmandade Santa Casa Misericórdia Marília
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50120915.1.0000.5413
Record Dates: First submitted 2016-07-02; First posted 2016-07-13 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Myocardial Infarction; Complications; Device, Vascular; Injury of Radial Artery; Injury; Blood Vessel, Femoral, Artery
Keywords: Vascular closure devices; Transradial approach; Transfemoral approach
MeSH Terms: conditions — Myocardial Infarction; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transradial approach (Active Comparator): Transradial approach primary percutaneous coronary intervention using the TR Band device to obtain hemostasis (n=125).
  Interventions: Procedure: Transradial primary percutaneous coronary intervention
- Transfemoral approach (Active Comparator): Transfemoral approach primary percutaneous coronary intervention using a vascular closure device to obtain hemostasis (n=125).
  Interventions: Procedure: Transfemoral primary percutaneous coronary intervention

INTERVENTIONS:
Procedure: Transradial primary percutaneous coronary intervention — Transradial coronary angiography will be performed by the Judkins technique using 6 French diameter sheaths and pre-molded catheters for selective catheterization of left and right coronary arteries. Primary percutaneous coronary intervention with stent deployment will be indicated when a culprit lesion is identified, with high probability of angiographic success, being ideally performed immediately after coronary angiography Procedures will be performed according to recommendations of current guidelines. To achieve hemostasis in the transradial approach, a radial compression device will be applied, to maintain patent antegrade flow.
  Arms: Transradial approach
Procedure: Transfemoral primary percutaneous coronary intervention — Transfemoral coronary angiography will be performed by the Judkins technique using 6 French diameter sheaths and pre-molded catheters for selective catheterization of left and right coronary arteries. Primary percutaneous coronary intervention with stent deployment will be indicated when a culprit lesion is identified, with high probability of angiographic success, being ideally performed immediately after coronary angiography Procedures will be performed according to recommendations of current guidelines. A vascular closure device will be used to achieve hemostasis in the transfemoral approach, preceded by systematic performance of femoral angiography and maintaining absolute bed rest for 60 minutes.
  Arms: Transfemoral approach

SUMMARY:
Primary percutaneous coronary intervention represents the gold standard for the treatment of ST-segment-elevation acute myocardial infarction. However, periprocedural bleedings are associated with an increased risk of mortality, re-infarction, and stroke. Although the prognostic value of access site related bleeding complications is still debated, transradial approach is associated with better short-term outcomes and reduced hospital stay as compared to transfemoral approach. The investigators aimed to compare transradial approach with transfemoral approach with systematic achievement of hemostasis by the implantation of a vascular closure device in a national multicentre randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* ST-segment elevation acute myocardial infarction patients during the first 12 hours of sympton onset;
* Intention to perform primary percutaneous coronary intervention;
* Signed informed consent;
* Patient eligible for transradial and transfemoral primary percutaneous coronary intervention, being pre-requisites: (a) familiarity of the operator with the radial and femoral techniques using vascular closure devices, (b) agreement of the operator to use the access route determined by the randomization process.

Exclusion Criteria:

* Less than 18 years of age;
* Pregnancy;
* Chronic use of vitamin K antagonists or direct thrombin inhibitors, or oral Xa-factor antagonists;
* Hypersensitivity to antiplatelet and/or anticoagulant drugs;
* Active bleeding or high bleeding risk (severe liver failure, active peptic ulcer, creatinine clearance < 30 mL/min, platelets count < 100.000 mm3);
* Uncontrolled systemic hypertension;
* Cardiogenic shock;
* Previous myocardial revascularization surgery with ≥ 1 internal mammary or radial artery graft;
* Documented chronic peripheral arterial disease preventing the use of the femoral technique;
* Severe concomitant disease with life expectancy below 12 months;
* Participation in drug or devices investigative clinical trials in the last 30 days;
* Medical, geographic or social conditions impairing the participation in the study or inability to understand and sign the informed consent term.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Major vascular access site complications | 48 hours post-procedure
  Major vascular complications related to arterial access site will be evaluated during hospitalization by physical examination and duplex ultrassonography and include major bleeding, retroperitoneal hemorrhage, compartment syndrome, pseudoaneurysm, arteriovenous fistula, limb ischemia or need for vascular surgery repair.

SECONDARY OUTCOMES:
Device success | 48 hours post-procedure
  The success of the device is defined as the attainment of adequate hemostasis at the end of the procedure, without the need to apply other compression methods.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro B Andrade, phD, Principal Investigator — Irmandade SCMM
Locations (1):
- Pedro Beraldo de Andrade, Marília, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Andrade PB, E Mattos LA, Tebet MA, Rinaldi FS, Esteves VC, Nogueira EF, Franca JI, de Andrade MV, Barbosa RA, Labrunie A, Abizaid AA, Sousa AG. Design and rationale of the AngioSeal versus the Radial approach In acute coronary SyndromE (ARISE) trial: a randomized comparison of a vascular closure device versus the radial approach to prevent vascular access site complications in non-ST-segment elevation acute coronary syndrome patients. Trials. 2013 Dec 18;14:435. doi: 10.1186/1745-6215-14-435. PMID 24345099